CLINICAL TRIAL: NCT01572259
Title: Assessment of the Role of the Growth Hormone (GH) Onthe Intestinal Triglyceride-rich-lipoproteins (TRL) Metabolism
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2011-001688-34; 2011-07 (Other: AP HM)
Record Dates: First submitted 2011-10-06; First posted 2012-04-06 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-08

CONDITIONS: Atherosclerotic Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis | interventions — Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- interruption of the growth hormone treatment. (Experimental)
  Interventions: Other: interruption of the traitment with growth hormone
- Patients traited by grouth hormone (Experimental)
  Interventions: Drug: Growth Hormone

INTERVENTIONS:
Drug: Growth Hormone
  Arms: Patients traited by grouth hormone
Other: interruption of the traitment with growth hormone
  Arms: interruption of the growth hormone treatment.

SUMMARY:
Atherosclerotic cardiovascular disease (ASCD) is the first cause of morbidity and mortality in insulin resistant states. The typical dyslipidemia that is associated with insulin resistance, which includes a postprandial increase of triglyceride-rich lipoproteins (TRL) with excess of intestinal triglyceride-rich-lipoprotein-apoB-48 (TRL-apoB-48), is felt to play an important role in the accelerated ASCD. Recently, intestinal TRL-apoB-48 overproduction appeared as a newly recognized component of insulin resistance. There is only a limited amount of information in the literature regarding the factors and the mechanisms modulating the metabolism of intestinal TRL-apoB-48 in the setting of insulin resistance

ELIGIBILITY:
Inclusion Criteria:

Male or feminine

* age from 18 to 70 years
* deficit in growth hormone informed by a peak lower than 10 mUI / l in answer to a test of hypoglycemia (or another test of stimulation if the hypoglycemia insulinique is dissuaded) (cf. attached the RCP of various growth hormone used at the adult)
* centre (treatments optimized previously will be maintained during all the duration of the study) thyréotrope, corticotrope and gonadotrope substituted well for at least 6 months
* IMC(CEREBRAL-MOTOR HANDICAPPED) < 30 kg / m2
* fasting blood glucose < 1,26 g/L
* clearance of the creatinine > 60 ml / min

Exclusion Criteria:

Nobody particularly protected: incapable major and private person of freedom, person hospitalized for another pathology; · nobody mastering the reading of the French language

* carrier patients of a tumor in service
* pregnant woman

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-09; Primary Completion 2016-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
To measure of Growth hormone | 3 YEARS
  that growth hormone modulates directly, or indirectly by the changes of insulin sensitivity

SECONDARY OUTCOMES:
to measure the adipocytokines levels (leptin, adiponectin, resistin) the metabolism (production and/or clearance) of the intestinal TRL | 3 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Maraninchi M, Calabrese A, Nogueira JP, Castinetti F, Mancini J, Mourre F, Pietri L, Benamo E, Albarel F, Morange I, Dupont-Roussel J, Nicolay A, Brue T, Beliard S, Valero R. Role of growth hormone in hepatic and intestinal triglyceride-rich lipoprotein metabolism. J Clin Lipidol. 2021 Sep-Oct;15(5):712-723. doi: 10.1016/j.jacl.2021.08.003. Epub 2021 Aug 16. PMID 34462238